CLINICAL TRIAL: NCT03220802
Title: Probiotic Modulation of Intestinal Microbiota in Long-term Intake of Proton Pump Inhibitors: Influence on Intestinal Inflammation and Digestion
Brief Title: Probiotic Modulation of Intestinal Microbiota in Long-term Intake of Proton Pump Inhibitors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Probiotics and PPI
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Patients on Long-term Proton Pump Inhibitor Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Test group (Experimental): participants receive a daily dose of OMNI-BiOTiC PPI for three months
  Interventions: Dietary Supplement: OMNI-BiOTiC PPI

INTERVENTIONS:
Dietary Supplement: OMNI-BiOTiC PPI — The study product consists of a sachet containing 4g of yellowish powder made of corn starch, maltodextrin, fructo-oligosaccharide P6, inulin P2, vegetable protein and 12 bacterial strains (Bacillus coagulans W183, Bacillus subtilus W201, Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Bifidobacterium lactis W51, Lactobacillus acidophilus W37, Lactobacillus acidophilus W22, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19, Propionibacterium freudenreichii W200, Lactobacillus rhamnosus W71, in a concentration of 2 x 109 cfu/g).

SUMMARY:
Long-term proton pump inhibitor use has been linked to intestinal dysbiosis, inflammation and gastrointestinal symptoms. Probiotics has been shown to correct dysbiosis, reduce inflammation and strengthen the gut barrier. The aim of this study is to evaluate the influence of a three months intervention with a probiotic on intestinal inflammation, bowel symptoms, dysbiosis and gut permeability.

DETAILED DESCRIPTION:
Proton pump inhibitors (PPIs) are among the top 5 most widely used drugs in the world. PPIs suppress the formation of gastric acid through the inhibition of hydrogen-potassium-adenosine-triphosphatase (H+ / K+ -ATPase) - a known proton pump in the parietal cells of the stomach. In practice, PPIs are commonly prescribed to treat GI disorders such as peptic ulcers and gastro-oesophageal reflux. They are also used prophylactically to prevent stress ulcers and to reduce GI toxicity associated with certain medications, including non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, and steroids, sometimes despite a paucity of evidence. PPI use has been associated with increased risk of enteric infections. A meta-analysis of 23 studies, comprising almost 300.000 patients, showed a 65% increase in the incidence of Clostridium difficile-associated diarrhoea among patients who used PPIs. Another meta-analysis of 11.280 patients, from six studies evaluating Salmonella, Campylobacter and other enteric infections, also found an increased risk due to acid suppression, with a greater association with PPI than with H2-receptor antagonists. Moreover, long term PPI use has been shown to be associated with bowel symptoms: A study from 2011 reported incidences of bloating, flatulence, abdominal pain and diarrhoea (43%, 17%, 7% and 2% of selected cases, respectively). In addition, PPIs are known to cause malabsorption of Vitamin B12 which may ultimately lead to Vitamin B12 deficiency. Very recently, PPI use was associated with an increase in mortality.

The gut microbiome plays an important role in enteric infections and bowel symptoms. The composition of the gut microbiome can inhibit or promote the microbial colonisation of the gut by microbial pathogens. Several mechanisms can influence bacterial growth or the immune system.

Long term PPI use is associated with profound changes in the gut microbiome. It is believed that these conditions are caused through the long-term suppression of gastric acid secretion (and thus shifting intragastric pH) which alters the natural habitat of resident microbiota. Furthermore, increased gastric pH might not sufficiently protect against oral or food-borne pathogens. We recently conducted a study at the Medical University of Graz where we could show that patients with long-term PPI therapy have dysbiosis associated with intestinal inflammation, increased gut permeability, bacterial translocation and systemic inflammation associated with a higher risk of complications and mortality in liver cirrhosis. (A. Horvath et al., Long-term proton pump inhibitor use increases intestinal dysbiosis, gut permeability, inflammation and mortality in patients with liver cirrhosis, UEG Journal, accepted) Probiotics are live microorganisms that have been demonstrated to alter gut flora and exhibit positive effects on numerous gastrointestinal complaints, strengthen the gut barrier and reduce inflammation parameters

We hypothesize that a three months probiotic intervention with OMNi BiOTiC PPI improves PPI induced dysbiosis, intestinal inflammation and gut permeability in patients on long term PPI therapy, leading to a decrease in bacterial translocation and a better gastrointestinal quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* willing to give written Informed Consent
* PPI intake for at least 6 months

Exclusion Criteria:

* Active infections at time of inclusion
* Antibiotic therapy within the last 14 days (includes prophylactic use)
* Inflammatory bowel diseases
* Consumption of pre/synbiotics other than the product provided during the trial
* Concomitant diseases or other circumstances that suggest that the patients are not eligible for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in faecal calprotectin levels due to the intervention | 6 months
  Calprotectin levels are measured in ng/mg stool using enzyme linked immunosorbent assay (ELISA) at baseline, after 3 months of intervention and after further 3 months of follow up

SECONDARY OUTCOMES:
changes in PPI associated Veillonella/Streptococcus dysbiosis index due to the intervention | 6 months
  relative abundance of bacteria in the gut microbiome will be assessed using 16S DNA sequencing, bacteria from the oral cavity will be especially investigated at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in faecal zonulin levels due to the intervention | 6 months
  Zonulin levels are measured in ng/mg stool using enzyme linked immunosorbent assay (ELISA) at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in serum endotoxin levels due to the intervention | 6 months
  endotoxin levels are measured in endotoxin units/ml serum using a cell based detection method at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in serum lipopolysaccharide binding protein (LBP) levels due to the intervention | 6 months
  LBP levels are measured in µg/ml serum using ELISA at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in serum sCD14 levels due to the intervention | 6 months
  sCD14 levels are measured in µg/ml serum using ELISA at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in serum VitB12 levels due to the intervention | 6 months
  VitB12 levels are measured as part of the routine laboratory report at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in health related quality of life due to the intervention | 6 months
  Quality of life will be described using the Short Form 36 Questionnaire at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in gastrointestinal quality of life due to the intervention | 6 months
  gastrointestinal quality of life will be described using the GIQLI questionnaire according to Eyparsch at baseline, after 3 months of intervention and after further 3 months of follow up
Changes in nutritional behaviour due to the intervention | 6 months
  Changes in nutritional behaviour due to the intervention will be determined by a food frequency questionnaire at baseline, after 3 months of intervention and after further 3 months of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No